CLINICAL TRIAL: NCT04686149
Title: Development of a Genome-based Platform to Predict Patients That Can Achieve Bladder Preservation After Preoperative Chemoradiotherapy in Muscle Invasive Bladder Cancer Patients
Brief Title: a Genome-based Platform to Predict Patients That Can Achieve Bladder Preservation in Muscle Invasive Bladder Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2020-1149
Record Dates: First submitted 2020-12-24; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Muscle-Invasive Bladder Carcinoma
Keywords: Bladder cancer; Bladder preservation; Genome-based platform; preoperative chemoradiotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — RNA sequencing was performed after RNA was isolated from the tissue sample obtained from TURB
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neo CCRT+Neo CTx +/- cystectomy: Patients receive neoadjuvant CCRT and neoadjuvant CTx. Radical cystectomy is performed depending on pathologic response. The patients showing clinical complete response after neoadjuvant CCRT and initially stage T2N0M0 are not treated with neoadjuvant chemotherapy.

SUMMARY:
This study is aimed to develop a genome-based platform to predict patients who can achieve bladder preservation after neoadjuvant treatment. The main treatments for invasive bladder cancer are radical cystectomy and intrapelvic lymph node dissection, but 50% of patients experience recurrence within 2 years after surgery. The recurrence after surgery is associate with T3 stage, the presence of invading soft tissue around the bladder and N1, lymph node metastasis. Therefore, various methods are being tried to reduce recurrence and metastasis, among which preoperative chemotherapy has been reported to increase survival rate. Based on this, preoperative chemotherapy followed by radical cystectomy are also recommended. However, there are several limitations; The surgery may be delayed in case of non-responsive to chemotherapy, the difficulty of tolerance of chemotherapy as the patients are relatively old in bladder cancer. Therefore, the preoperative concurrent chemoradiotherapy can be considered as a treatment effectively lower the recurrence. In several retrospective study has reported that preoperative radiation induces the down-staging and leads to prolonged progression free survival. However, after radical cystectomy, there is discomfort for patients regarding the removal of the bladder. Treating the bladder while preserving the bladder is getting its attention. The representative treatment is performing neoadjuvant concurrent chemotherapy followed by transurethral resection of bladder tumor. The bladder preserving treatment is performed in patients who have unresectable, locally advanced bladder cancer or are not medically appropriate for surgery. The 5-year overall survival is reported to be around 50-60%. To date, no clinical trial has been conducted to compare whether concurrent chemoradiotherapy can achieve the comparable clinical outcome as radical cystectomy in operable conditions. Therefore, in order to perform the bladder preserving treatment, a platform selecting patients who can preserve the bladder from bladder preserving treatment in advance is needed. Responsiveness to radiotherapy is a combination of various factors, and radiation sensitivity of tumors is the most important. The recent study has been demonstrated that physician can predict radiation sensitivity using genomic data. In this study, we intend to develop a platform that can predict responsiveness to radiotherapy and select patients who can preserve bladder using genomic information.

DETAILED DESCRIPTION:
The treatment in this study is one of the standard treatments suggested by the NCCN guidelines. Bladder is preserved when neoadjuvant concurrent chemoradiotherapy is performed after transurethral resection of bladder tumor and complete remission is achieved through the cystoscopy. If complete response is not achieved, additional chemotherapy is performed. In case that complete response is not achieved through the cystoscopy after additional chemotherapy, cystectomy is performed. If complete response is achieved, the bladder is preserved.

Before treatment, the following are obtained; Medical history and physical examination, Tissue acquisition through transurethral resection of bladder tumor, Blood Test (CBC), Chemistry Test (SMA), staging through pelvic CT or MRI, cystoscopy, PET-CT or chest CT.

Cisplatin based concurrent chemoradiotherapy is conducted 4 times during the radiotherapy. AFter radiotherapy, the gemcitabine/cisplatin or gemcitabine/carboplatin treatment is performed. The target delineation is performed in 3mm simulation CT for radiotherapy. To consider the uncertainty of breath, the 4D CT is taken. GTV includes primary lesions and lymph node based on diagnostic CT, MRI, and PET-CT. CTV covers the entire bladder with microscopic margin of GTV. PTV1 is defined as extending 1.5cm from the entire bladder. PTV2 is defined as extending 1.5cm from GTV. Radiotherapy is performed using 3D conformal radiotherapy, intensity-modulated radiotherapy, volumetric modulated Arc therapy. Radiotherapy is administered daily, five times a week according to the NCCN guidelines. Each treatment is performed with bladder empty. radiotherapy is performed 20 fractions in total. For the first 15 fractions, 2.65Gy administered for PTV1 including the entire bladder. For rest 5 fractions, 3 Gy for PTV2 is administered. Totally, 55 Gy is administered.

If complete response is not achieved, the surgery and timing of surgery are determined by the urologist according to the location and severity of the primary cancer. The biopsy if performed using cystoscopy. If the findings are complete response, no additional treatment is performed, and if not, radical cystectomy is performed.

The treatment response is evaluated based on standard treatment process. During the treatment, the regular check up is conducted to evaluate the acute toxicity regarding treatment. After bladder preserving treatment, the pelvic CT, MRI and cystoscopy is used for evaluation.

The acquired specimens are ;used for RNA sequencing and organoid construction. The RNA sequencing is used to analyze the differentially expressed based on treatment response to neoadjuvant concurrent chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 19 years old
2. Clinically or histologically diagnosed urothelial carcinoma bladder cancer
3. Patients who satisfy all of the following conditions with bladder cancer stage T2-4a, N0-1 according to 8th edition of American Joint Committee on Cancer

   * Muscle invasive bladder cancer confirmed by cystoscopy
   * Stage T2-4a, N0-1 in CT or MRI
4. Performance status 0 or 1 based on ECOG
5. Patients agreed to provide the tissue sample obtained from TURB
6. Diseases can be evaluated according to RECIST Version 1.1
7. Patients who voluntarily agreed to informed consent

Exclusion Criteria:

1. Patients with distant metastasis
2. Patients with uncontrolled viral infection (HIV, HBV, HCV)
3. Patient who are pregnant, or have possibility of pregnancy and are on lactating
4. Hypersensitivity or history of allergic to the drug being used
5. Patients with cerebrovascular disease, complications, and infections that are not medically controlled
6. Patients with history of other malignant diseases within the past 5 years (excluding cured non-melanoma skin cancer or in situ cervical cancer)
7. Those who are taking drugs that can cause drug interactions with chemotherapy
8. Patients who withdraw consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with muscle invasive bladder cancer are subject to this trial. For bladder preservation, the patients receive neoadjvuvant CCRT. In case that clinical CR status obtained after CCRT in patients initally T2N0M0, no additional treatment is performed. Patients without clinical CR status are treated with neoadjuvant chemotherapy. After chemotherapy, the response is evaluated. If residual tumor is found, the radical cystectomy is performed.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Bladder preservation rate | up to 2 years
  The rate of patients achieve bladder preservation without radical cystectomy

SECONDARY OUTCOMES:
Pathologic complete response rate | up to 2 years
  The rate of lesions detected as pathologically complete response after neoadjuvant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Woong Sub Koom, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Research related documents will be stored in a file with a separate password under the responsibility of the lead researcher and stored in a locked laboratory. These research-related records will be kept for 3 years from the time the research is completed, and after that, the research team will discard the documents.
  Tissue samples obtained from patients are subjected to genome analysis by extracting RNA and DNA. Patient registration information is encrypted and stored separately, and stored in freezer at -80°C until experimentation at Yonsei University Medical Research Institute under the supervision of the research director.